CLINICAL TRIAL: NCT06940349
Title: A Phase 1b/2 Open Label, Dose Escalating, Single Center Study to Evaluate the Safety, Tolerability and Initial Efficacy of Palbociclib + Sunitinib Oral Kinase Inhibitor Combination as a Treatment for Advanced Solid Tumors
Brief Title: Interventional Study to Evaluate the Combination of Palbociclib + Sunitinib as a Treatment for Advanced Solid Tumors
Acronym: COPS-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Idit Peretz, Principal Investigator, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104420-RMC
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors Refractory to Standard Therapy
Keywords: COPS study; phase 1/phase 2 study; combination Palbociclib and Sutent
MeSH Terms: interventions — palbociclib; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Palbociclib and Sunitinib combination (Experimental): All patients will be administered Sunitinib (S) 25 mg + Palbociclib (P) 75 mg, both once daily for 5 consecutive days and 2 days off schedule for the first week and then the dose can be escalated to S 37.5 mg + P 75 mg, Both once daily for 5 consecutive days and 2 days off schedule per week. From the second week onwards, dose can be escalated to S 37.5 mg + P 75 mg, Both once daily for 7 consecutive days, per physician discretion.
  Interventions: Drug: Palbociclib; Drug: Sunitinib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib and Sunitinib
Drug: Sunitinib — Palbociclib and Sunitinib

SUMMARY:
The goal of this clinical trial is to learn if a combination of Palbociclib and Sunitinib is safe and effective in various solid tumors.

The main questions it aims to answer are:

* Is the drugs combination safe for the participants?
* Is the drug combination effective in all solid malignancies? It is a single arm study, phase 1b/2, dose escalation and expansion, to determine the safety, tolerability and initial efficacy of this combination.

Participants will:

* Take the drugs combination every day for 5 executive days, and 2 days of, in a 28 days cycle, for up to a year.
* Visit the clinic once every 2 weeks for checkups and tests

DETAILED DESCRIPTION:
Based on the observed in vivo synergistic effects of the Palbociclib and Sunitinib combination on human tumor growth in the PDX models, and the expectation that major pharmacodynamic interactions are not expected, the Investigator initiated a Phase 1b/2 study to evaluate the safety, tolerability and initial efficacy of Palbociclib + Sunitinib oral kinase inhibitor combination as a treatment for advanced solid tumors.

The study population will include 20-100 patients with documented Stage IV, incurable/refractory metastatic solid tumors of the following types whom have failed at least one standard course of therapy: (1) Gastric adenocarcinoma, (2) Ovarian Epithelial, Fallopian Tube, and Primary Peritoneal cancer (FIGO classification), (3) Breast cancer, (4) NSCLC, (5) Colorectal cancer, (6) Cholangiocarcinoma, (7) Pancreatic cancer and (8) Carcinosarcoma, any tissue origin.

(9) High grade Neuroendocrine Carcinoma, from any tissue origin. (10) Sarcoma, all histological types. (11) Any other solid tumor.

All patients will be administered 25 mg S:75 mg P, both once daily for 5 consecutive days and 2 days off schedule for the first week and then the dose can be escalated to 37.5 mg S:75 mg P, Both once daily for 5 consecutive days and 2 days off schedule per week. From the second week onwards, dose can be escalated to 37.5 mg S:75 mg P, Both once daily for 7 consecutive days, per physician discretion. Sunitinib dose will be evaluated in each clinic visit, dose can be adjusted to alternately 37.5mg/25mg or be reduced to 25 mg daily, by patient tolerance and adverse events.

Both drugs will be administered by mouth, taken together with food

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with Stage IV incurable/refractory metastatic solid tumors or locally advanced incurable/refractory tumor, who have one of the following tumor types:

  (1) Gastric adenocarcinoma, (2) Ovarian Epithelial, Fallopian Tube, and Primary Peritoneal cancer (FIGO classification), (3) Breast cancer, (4) NSCLC, (5) Colorectal cancer, (6) Cholangiocarcinoma, (7) Pancreatic cancer, (8) Carcinosarcoma (any tissue origin), (9) High grade Neuroendocrine Carcinoma, from any tissue origin, (10) Sarcoma, all histological types, (11) Any other solid tumor.
* Patients who have failed all other appropriate lines of therapy or who have refused treatment(s) of choice
* Life expectancy of greater than 8 weeks
* Clinical performance status of ECOG 0-2
* Able to understand and sign the Informed Consent Form
* Must be able to adhere to the study visit schedule and other protocol requirements.

Hematology criteria:

Absolute neutrophils count greater than 1000/mm3 without support of filgrastim Normal WBC (>3000/mm3). Hemoglobin greater than 8.0 g/dL Platelet count greater than 80,000/mm3

* Serology:
* Seronegative for HIV antibody
* Documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test
* Patients with active HBV must have:
* HBV DNA < 500 IU/mL obtained within 28 days prior to initiation of study treatment
* received anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study
* Patients with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV
* Chemistry:
* Serum ALT/AST less than three times the upper limit of normal (ULN)/ less than five times ULN if liver metastasis present
* Serum creatinine less than or equal to 1.6 mg/dL
* Total bilirubin no more than x1.5 times the ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dL.
* Non-pregnant (via negative pregnancy test)/non-breast-feeding women and women with no intention to become pregnant/to breast-feed during the term of the trial and for at least three months after cessation of the P+S treatment
* More than 14 days must have elapsed since any prior systemic therapy before day 1, and patients' toxicities must have recovered to a Grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures, local radiotherapy with the past two weeks, as long as all toxicities have recovered to Grade 1 or less.

Exclusion Criteria:

* Inclusion Criteria:

  * Age ≥18 years
  * Patients with Stage IV incurable/refractory metastatic solid tumors or locally advanced incurable/refractory tumor, who have one of the following tumor types:

    (1) Gastric adenocarcinoma, (2) Ovarian Epithelial, Fallopian Tube, and Primary Peritoneal cancer (FIGO classification), (3) Breast cancer, (4) NSCLC, (5) Colorectal cancer, (6) Cholangiocarcinoma, (7) Pancreatic cancer, (8) Carcinosarcoma (any tissue origin), (9) High grade Neuroendocrine Carcinoma, from any tissue origin, (10) Sarcoma, all histological types, (11) Any other solid tumor.
  * Patients who have failed all other appropriate lines of therapy or who have refused treatment(s) of choice
  * Life expectancy of greater than 8 weeks
  * Clinical performance status of ECOG 0-2
  * Able to understand and sign the Informed Consent Form
  * Must be able to adhere to the study visit schedule and other protocol requirements
  * Hematology:
* Absolute neutrophils count greater than 1000/mm3 without support of filgrastim
* Normal WBC (>3000/mm3).
* Hemoglobin greater than 8.0 g/dL
* Platelet count greater than 80,000/mm3

  • Serology:
* Seronegative for HIV antibody
* Documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test
* Patients with active HBV must have:
* HBV DNA < 500 IU/mL obtained within 28 days prior to initiation of study treatment
* received anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study
* Patients with a history of HCV infection but who are negative for HCV RNA by PCR will be considered non-infected with HCV

  • Chemistry:
* Serum ALT/AST less than three times the upper limit of normal (ULN)/ less than five times ULN if liver metastasis present
* Serum creatinine less than or equal to 1.6 mg/dL
* Total bilirubin no more than x1.5 times the ULN, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dL.

  * Non-pregnant (via negative pregnancy test)/non-breast-feeding women and women with no intention to become pregnant/to breast-feed during the term of the trial and for at least three months after cessation of the P+S treatment
  * More than 14 days must have elapsed since any prior systemic therapy before day 1, and patients' toxicities must have recovered to a Grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures, local radiotherapy with the past two weeks, as long as all toxicities have recovered to Grade 1 or less.

Exclusion Criteria:

* Known active current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections (including but not limited to tuberculosis, atypical mycobacterial disease, and herpes zoster), human immunodeficiency virus (HIV), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) or oral antibiotics within 1 week of day 1
* History of severe immediate hypersensitivity reaction to any of the agents used in this study
* Uncontrolled hypertension
* Proteinuria >3 grams per day
* Subjects who have received any investigational drug or used investigational device within two weeks preceding screening
* Active consumption of illicit drugs within one month preceding screening
* Serious psychiatric or psychological disorders
* Patients with significant cardiac, respiratory or active malignancy disease comorbidities.
* Women of child-bearing potential who intend to become pregnant or breast-feed or who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Primary safety analysis | To be assessed every Disease Monitoring and Safety Board, Every 4 months.
  To evaluate the incidence and severity of treatment related adverse events of the Palbociclib and Sunitinib combination using CTCAE v5.0 in all indications
Primary efficacy analysis | Through study completion, estimated 18 months.
  To determine the percentage of Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progression of Disease (PD) via RECIST criteria, based on the results of the imaging studies. Imaging studies will be carried out at Screening and every two months after treatment initiation.

SECONDARY OUTCOMES:
Response rate | Through study completion, estimated 18 months.
  To determine the response rate (sum of Complete Response (CR) + Partial Response (PR) for all patients with all indications
Time to progression | Through study completion, estimated 18 months.
  To determine the Time-To-Progression (TTP) for all patients with all indications
Progression free survival | Through study completion, estimated 18 months.
  To determine the Progression-Free Survival (PFS) for all patients with all indications
Quality of life by EORTC validated questionnaires in all indications, and disease specific indications | Through study completion, estimated 18 months.
  To assess the Quality of Life (QoL) via disease-specific questionnaires for all patients with all indications

CONTACTS AND LOCATIONS:
Overall Officials: idit Peretz, MD,MBA, Principal Investigator — Rabin Medical Center
Locations (1):
- Davidoff cancer center, RMC, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No